CLINICAL TRIAL: NCT04080882
Title: A Multicenter, Randomized, Dose-Ranging, Double-Blind, Placebo-Controlled Study to Evaluate Safety and Efficacy of AbobotulinumtoxinA for the Treatment of Moderate to Severe Platysmal Bands
Brief Title: Safety and Efficacy of AbobotulinumtoxinA for the Treatment of Platysmal Bands
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 43USD1804
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2021-01

CONDITIONS: Platysmal Bands

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AbobotulinumtoxinA dose 1 (Active Comparator): AbobotulinumtoxinA dose 1 injected into platysma bands
  Interventions: Biological: AbobotulinumtoxinA dose 1
- placebo (Placebo Comparator): placebo injected into platysma bands
  Interventions: Other: Placebo
- AbobotulinumtoxinA dose 2 (Active Comparator): AbobotulinumtoxinA dose 2 injected into platysma bands
  Interventions: Biological: AbobotulinumtoxinA dose 2
- AbobotulinumtoxinA dose 3 (Active Comparator): AbobotulinumtoxinA dose 3 injected into platysma bands
  Interventions: Biological: AbobotulinumtoxinA dose 3

INTERVENTIONS:
Biological: AbobotulinumtoxinA dose 1 — Treatment of platysmal bands
  Arms: AbobotulinumtoxinA dose 1
Other: Placebo — Treatment of platysmal bands
  Arms: placebo
Biological: AbobotulinumtoxinA dose 2 — Treatment of platysmal bands
  Arms: AbobotulinumtoxinA dose 2
Biological: AbobotulinumtoxinA dose 3 — Treatment of platysmal bands
  Arms: AbobotulinumtoxinA dose 3

SUMMARY:
Interventional phase 2 study to evaluate safety and efficacy of abobotulinumtoxinA for the treatment of platysmal bands.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe platysmal bands at maximum contraction as assessed by the Investigator using a photographic scale
* Platysmal bands graded as Level 3 or 4 at maximum contraction as assessed by the subject using a photographic scale

Exclusion Criteria:

* Botulinum toxin treatment of any serotype below the lower orbital rim, in the neck or chest within 12 months prior to study treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Galderma Research Site, Encinitas, California
  - Galderma Research Site, Encino, California
  - Galderma Research Site, Boynton Beach, Florida
  - Galderma Research Site, Miami, Florida
  - Galderma Research Site, New Orleans, Louisiana
  - Galderma Research Site, Baltimore, Maryland
  - Galderma Research Site, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | AbobotulinumtoxinA Dose 1
Started | 20 | 60
Completed | 18 | 58
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: Due to business decision study did not proceed to enroll dose 2 or dose 3.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AbobotulinumtoxinA Dose 1 | Total
Number analyzed (Participants) | 20 | 60 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 60 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (8.56) | 52.1 (7.74) | 51.7 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 58 | 78
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 11 | 14
  Not Hispanic or Latino | 17 | 49 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 18 | 57 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 60 | 80
Fitzpatrick Skin Type (FST) [Count of Participants; unit: Participants] — FST I: white; very fair; red or blond hair; blue eyes; freckles. always burns, never tans.
  FST II: white; fair; red or blond hair; blue, hazel or green eyes. usually burns, tans with difficulty.
  FST III: cream white; fair with any eye or hair color; very common. sometimes mild burn, gradually tans.
  FST IV: brown; typical Mediterranean Caucasian skin. rarely burns, tans with ease.
  FST V: dark brown; Middle Eastern skin types. very rarely burns, tans very easily.
  FST VI: Skin color - black. Skin Characteristics - never burns, tans very easily.
  Participants
    FST I | 0 | 0 | 0
    FST II | 9 | 17 | 26
    FST III | 5 | 25 | 30
    FST IV | 4 | 15 | 19
    FST V | 1 | 1 | 2
    FST VI | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate at Month 1 for a Single Dose of abobotulinumtoxinA Compared to Placebo
Description: A responder is defined as a subject who achieves grade 1 or 2 in platysmal band severity on the Investigator Live Assessment (ILA).
Time Frame: Month 1 after treatment
Population: Due to business decision study did not proceed to enroll dose 2 or dose 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AbobotulinumtoxinA Dose 1
Number analyzed (Participants) | 20 | 60
Participants | 3 | 36

ADVERSE EVENTS:
Time Frame: 5 months
Description: Due to business decision study did not proceed to enroll dose 2 or dose 3.
Arm/Group | Placebo | AbobotulinumtoxinA Dose 1
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/60
Other Adverse Events (participants affected / at risk) | 7/20 | 14/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | AbobotulinumtoxinA Dose 1 (N=60)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 5 (5)
Injection site heamorrhage (General disorders) | 0 (0) | 3 (3)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Viral upper respiratory tract infectinon (Infections and infestations) | 1 (1) | 2 (3)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agree not to present or publish any data or reports collected individually or by subgroup of sites prior to full, initial publication based on all data obtained from all sites.

DOCUMENTS (2):
  • Study Protocol (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT04080882/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT04080882/SAP_001.pdf